CLINICAL TRIAL: NCT02546986
Title: A Phase 2 Multicenter, Randomized, Placebo Controlled, Double Blind Study to Assess the Safety and Efficacy of CC-486 (Oral Azacitidine) in Combination With Pembrolizumab (MK-3475) Versus Pembrolizumab Plus Placebo in Subjects With Previously Treated Locally Advanced or Metastatic Non-small Cell Lung Cancer
Brief Title: Safety and Efficacy Study of CC-486 With MK-3475 to Treat Locally Advanced or Metastatic Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CC-486-NSCL-001
Expanded Access: NCT03723135 (Approved for marketing)
Record Dates: First submitted 2015-08-20; First posted 2015-09-11 (Estimated); Results first posted 2018-05-14 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-07

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: CC-486; Azacitidine; Oral azacitidine; Methyltransferase inhibitor; Hypomethylation; Hypomethylating agent; Epigenetic; MK-3475; Pembrolizumab; Keytruda; PD-1; PD-L1; ImmunotherapyAdvanced non-small cell lung cancer; Metastatic non-small cell lung cancer; Non-small cell lung cancer; NSCLC; Merck Pembrolizumab (Keynote-117)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — cc-486; Azacitidine; pembrolizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CC-486 plus Pembrolizumab (Experimental): In the experimental arm, participants will receive a combination of two investigational drugs, CC-486 and pembrolizumab every 21-days.
  Interventions: Drug: CC-486; Drug: Pembrolizumab
- Pembrolizumab plus Placebo (Experimental): In this control arm, participants will receive pembrolizumab as a 30 minute IV infusion on day 1 of each 21-day cycle and placebo will be administered by mouth daily on days 1 to 14 of each 21 day cycle. Placebo will also be administered in order to allow blinding of the study.
  Interventions: Drug: Pembrolizumab; Drug: Placebo

INTERVENTIONS:
Drug: CC-486 — CC-486 will be administered orally at a dose of 300 mg daily on days 1-14 of each 21-day cycle.
  Other Names: Oral Azacitidine
  Arms: CC-486 plus Pembrolizumab
Drug: Pembrolizumab — Pembrolizumab will be administered as a 30-minute IV infusion on day 1 of each 21-day cycle.
  Other Names: MK-3475
Drug: Placebo — Placebo will be administered orally daily on days 1-14 of each 21-day cycle.
  Arms: Pembrolizumab plus Placebo

SUMMARY:
The purpose of this study is to determine whether the combination therapy of CC-486 (oral azacitidine) and pembrolizumab provides improved patient outcomes compared to pembrolizumab alone in patients with previously treated locally advanced or metastatic non-small cell lung cancer.

DETAILED DESCRIPTION:
This is a Phase 2, multicenter, international, randomized, placebo controlled, double-blind study to assess the safety and efficacy of CC-486 and pembrolizumab combination therapy versus pembrolizumab plus placebo in previously treated patients with locally advanced or metastatic non-small cell lung cancer (NSCLC) who had received one prior platinum-based chemotherapy regimen.

Approximately 100 participants will be randomized 1:1 to receive CC-486 plus pembrolizumab or placebo plus pembrolizumab as follows:

* Arm A: CC-486 300 mg administered orally daily on days 1 to 14 plus pembrolizumab 200 mg administered as a 30-minute IV infusion on day 1 of a 21-day cycle
* Arm B: Placebo administered orally daily on days 1-14 plus pembrolizumab 200 mg administered as a 30-minute IV infusion on day 1 of a 21-day cycle

Randomization will be stratified between treatment arms by histology (non-squamous versus squamous).

The decision to discontinue a patient, which will not be delayed or refused by the Sponsor, remains the responsibility of the treating physician. However, prior to discontinuing a patient, the Investigator may contact the medical monitor and forward appropriate supporting documents for review and discussion.

In the follow-up phase, anticancer treatment administered following the last dose of investigational product (IP) and survival will be followed every 8 weeks until death, withdrawal of consent, or lost-to follow-up, whichever occurs first, or the End of Trial.

The study will be conducted in compliance with the International Council on Harmonisation (ICH) of Technical Requirements for Registration of Pharmaceuticals for Human Use/Good Clinical Practice (GCP) and applicable regulatory requirements.

Primary analysis will be conducted when 70 Progression Free Survival (PFS) events have occurred.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is ≥ 18 years of age at the time of signing the informed consent form.
2. Participant has histologically or cytologically confirmed squamous or non-squamous non-small cell lung cancer (NSCLC).
3. Participant has stage IIIB or IV NSCLC (American Joint Committee on Cancer [AJCC] Staging Manual, 7th edition [Edge, 2009]) and was pretreated with only 1 prior systemic platinum based chemotherapy.
4. Participant has provided a formalin fixed tumor tissue sample from a biopsy of a tumor lesion either at the time of or after the diagnosis of metastatic disease has been made and from a site not previously irradiated to assess for a protein known as Programmed death-ligand 1( PD-L1) status. Fine needle aspirates, endobronchial ultrasound (EBUS) or cell blocks are not acceptable. Needle or excisional biopsies, or resected tissue is required. Archival tissue may be acceptable. Submission of formalin-fixed paraffin embedded tumor tissue sample blocks are preferred; if submitting unstained slides, the slides should be freshly cut and submitted to the testing laboratory within 14 days from site slide sectioning date otherwise a new specimen will be requested.
5. Participant has radiographically-documented measurable disease, as per Response Evaluation Criteria In Solid Tumors version 1.1 (RECIST v1.1).
6. Particiapant has an Eastern Cancer Oncology Group (ECOG) performance status of 0 to 1.
7. Participant has adequate organ functions, evidenced by the following:

   1. Aspartate aminotransferase (AST), Serum glutamic oxaloacetic transaminase (SGOT), alanine aminotransferase (ALT), serum glutamic pyruvic transaminase (SGPT) ≤ 2.5 x upper limit of normal range (ULN), or ≤ 5 x ULN range if liver metastasis present
   2. Total bilirubin ≤ 1.5 x ULN
   3. Serum creatinine ≤ 1.5 x ULN
   4. Potassium within normal range, or correctable with supplements
8. Participant has adequate bone marrow function, evidenced by the following:

   1. Absolute neutrophil count ≥ 1.5 x 10^9 cells/L
   2. Platelets ≥ 100 x 10^9 cells/L
   3. Hemoglobin ≥ 9 g/dL
   4. International normalized ratio (INR) or prothrombin time (PT) ≤ 1.5 x ULN unless participant is receiving anticoagulant therapy as long as prothrombin time (PT) or partial thromboplastin time (PTT) is within therapeutic range of intended use of anticoagulants
   5. Activated partial thromboplastin time (aPTT) ≤ 1.5 x ULN unless participant is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
9. Female of childbearing potential (FCBP) (defined as a sexually mature woman who 1) has not undergone a hysterectomy (the surgical removal of the uterus) or bilateral oophorectomy (the surgical removal of both ovaries) or, 2) if ≥ 45 years old has not been naturally postmenopausal for at least 24 consecutive months (ie, has had menses at any time during the preceding 24 consecutive months) must:

   1. Have two negative pregnancy tests as verified by the Investigator prior to starting study therapy. She must agree to ongoing pregnancy testing during the course of the study, and after end of study treatment. This applies even if the participant practices true abstinence* from heterosexual contact.
   2. Either commit to true abstinence* from heterosexual contact (which must be reviewed on a monthly basis) or agree to use, and be able to comply with two effective methods of contraception without interruption, 28 days prior to starting IP, during the study therapy (including dose interruptions), and for 120 days after discontinuation (or longer if required by local requirements) of study therapy. The two methods of contraception can either be two barrier methods or a barrier method plus a hormonal method to prevent pregnancy.
10. Male participants must practice true abstinence* (which must be reviewed on a monthly basis) or agree to the use a condom during sexual contact with a pregnant female or a female of childbearing potential while participating in the study, during dose interruptions and for at least 3 months following investigational product discontinuation (or longer if required by local requirements), even if he has undergone a successful vasectomy.

    * True abstinence is acceptable when this is in line with the preferred and usual lifestyle of the participant. Note: Periodic abstinence (eg, calendar, ovulation, symptothermal, postovulation methods) and withdrawal are not acceptable methods of contraception.
11. Participant is willing to adhere to the study visit schedule and other protocol requirements.
12. Participant understands and voluntarily signs an informed consent document prior to any study related assessments or procedures are conducted.

Exclusion Criteria:

1. Participants with non-squamous histology has known or unknown sensitizing epidermal growth factor receptor (EGFR) and/or anaplastic lymphoma kinase positive (ALK) mutation. Note: Participants with squamous histology and unknown EGFR and ALK mutational status are eligible.
2. Participant has received more than one line of therapy for stage IIIB or IV disease
3. Participant has been previously treated with azacitidine (any formulation), decitabine, or any other hypomethylating agent.
4. Particpant has received prior therapy with any other anti-PD-1, or PD-L1 or PD-L2 agent or an antibody targeting other immuno-regulatory receptors or mechanism, including participation in any other pembrolizumab trial and treatment with pembrolizumab.

   a. Examples of such antibodies include (but are not limited to) antibodies against indoleamine 2,3-dioxygenase (IDO), PD-L1, IL-2R, glucocorticoid-induced tumor necrosis factor receptor (GITR).
5. Participant has had a prior monoclonal antibody within 4 weeks prior to study Day 1 or who has not recovered (i.e. ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
6. Participant is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks prior to administration of pembrolizumab and CC-486
7. Participant has previous severe hypersensitivity reaction to another monoclonal antibody (mAb).
8. Participant has a known or suspected hypersensitivity to azacitidine, mannitol, or any other ingredient used in the manufacture of CC-486 (see the Azacitidine IB).
9. Participant has had radiotherapy ≤ 4 weeks or limited field radiation for palliation
10. Participant has received radiation therapy to the lung that is > 30 Gy within 6 months of the first dose of trial treatment
11. Participant has received a live-virus vaccination within 30 days of planned treatment start. Seasonal flu vaccines that do not contain live virus are permitted.
12. Participant has not recovered from the acute toxic effects of prior anticancer therapy, radiation, or major surgery/significant trauma.
13. Participant has an active infection requiring therapy.
14. Participant has had an allogenetic tissue/solid organ ransplant.
15. Participant has active autoimmune disease that has required systemic treatment within the past 2 years (eg, with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
16. Participant has known active Hepatitis B, Hepatitis C or tuberculosis. Active Hepatitis B is defined as a known positive HBsAg result. Active Hepatitis C is defined by a known positive Hepatitis C antibody result and known quantitative Hepatitis C virus (HCV) ribonucleic acid (RNA) results greater than the lower limits of detection of the assay.
17. Participant has had any other malignancy within 5 years prior to randomization, with the exception of adequately treated in situ carcinoma of the cervix, uterus, or nonmelanomatous skin cancer (all treatment of which should have been completed 6 months prior to enrollment).
18. Participant has a history of inflammatory bowel disease (eg, Crohn's disease, ulcerative colitis), celiac disease (ie, sprue), prior gastrectomy or upper bowel removal, or any other gastrointestinal disorder or defect that would interfere with the absorption, distribution, metabolism, or excretion of the IP and/or predispose the participant to an increased risk of gastrointestinal toxicity.
19. Participant has persistent diarrhea or clinically significant malabsorption syndrome or known sub-acute bowel obstruction ≥ Grade 2, despite medical management
20. Participant has significant active cardiac disease within the previous 6 months including unstable angina or angina requiring surgical or medical intervention, significant cardiac arrhythmia, or New York Heart Association (NYHA) class 3 or 4 congestive heart failure.
21. Participant has history of interstitial lung disease (ILD) OR a history of pneumonitis that has required oral or IV steroids. Participants whose pneumonitis was solely as a result of radiation therapy for their NSCLC would not be excluded from the study unless they received oral/IV steroids to manage the pneumonitis.
22. Participant has a known history or current diagnosis of human immunodeficiency virus (HIV) infection, regardless of treatment status.
23. Participant has any other concurrent severe and/or uncontrolled medical condition that would, in the Investigator's judgment, contraindicate patient participation in the clinical study (eg, chronic pancreatitis, etc.).
24. Participant with uncontrolled or symptomatic central nervous system (CNS) metastases and/or carcinomatous meningitis Participants with controlled and asymptomatic CNS metastases may participate in this trial. The patient must have completed any prior treatment for CNS metastases (must include radiotherapy and/or surgery) ≥ 28 days (≥ 14 days for stereotactic radiosurgery) and, if on corticosteroid therapy, should be receiving a stable dose of no greater than 4 mg/d dexamethasone (or equivalent anti-inflammatory potency of another corticosteroid) for at least 14 days before start of study treatment). Patients must not be receiving corticosteroids for brain metastases.
25. Partcipant has not recovered from the acute toxic effects (Common Terminology Criteria for Adverse Events [CTCAE] grade ≤ 1) of prior anticancer therapy, radiation, or major surgery/significant trauma (except alopecia or other toxicities not considered a safety risk for the particiapants at the Investigator's discretion).
26. Participant has an impaired ability to swallow oral medication.
27. Participant is pregnant or breast feeding.
28. Participant has any condition that confounds the ability to interpret data from the study.
29. Participant is or has an immediate family member (spouse or children) who is investigational site or sponsor staff directly involved with this trial, unless prospective Institutional Review Board (IRB) approval (by chair or designee) is given allowing exception to this criterion for a specific participant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-10-09 (Actual); Primary Completion 2017-04-13 (Actual); Study Completion 2025-07-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (33):
- United States (10):
  - Palo Verde Hematology Oncology, Glendale, Arizona
  - UCLA Hematology Oncology, Los Angeles, California
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - University Cancer and Blood Center, LLC, Athens, Georgia
  - Research Medical Center, Kansas City, Missouri
  - Washington Univ School of Medicine, St Louis, Missouri
  - North Shore Hematology Oncology Associates, East Setauket, New York
  - Local Institution - 006, New York, New York
  - NYU Langone Medical Center, New York, New York
  - Vanderbilt Univ Medical Center, Nashville, Tennessee
- France (4):
  - Local Institution - 204, Lyon
  - Local Institution - 200, Marseille
  - Local Institution - 203, Toulouse
  - Local Institution - 201, Villejuif
- Germany (4):
  - Local Institution - 302, Berlin
  - Local Institution - 304, Cologne
  - Local Institution - 300, Esslingen am Neckar
  - Local Institution - 301, Löwenstein
- Local Institution - 903, Athens, Greece
- Italy (7):
  - Local Institution - 601, Aviano
  - Local Institution - 604, Catania
  - Local Institution - 602, Milan
  - Local Institution - 606, Milan
  - Local Institution - 603, Napoli, Campania
  - Local Institution - 600, Novara
  - Local Institution - 605, Roma
- Spain (7):
  - Local Institution - 705, Barakaldo
  - Local Institution - 702, Barcelona
  - Local Institution - 703, Madrid
  - Local Institution - 701, Madrid
  - Local Institution - 704, Madrid
  - Local Institution - 706, Madrid
  - Local Institution - 700, Valencia

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSClinicalTrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was a multicenter study with 25 sites from the United States, France. Germany, Italy, and Spain.
Pre-assignment Details: Qualified participants were randomized in a 1:1 ratio to one of the two treatment groups. Randomization was stratified by cancer histology (non-squamous versus squamous).
Groups:
- CC-486 and Pembrolizumab (CC-486 + PBZ): Participants received CC-486 300 mg tablets by mouth (PO) on Days 1-14 of each 21-day treatment cycle and pembrolizumab (PBZ) 200 mg administered as a 30-minute intravenous (IV) infusion on Day 1 of each 21-day cycle until radiologic disease progression (DP), unacceptable toxicity, initiation of a new anticancer therapy, withdrawal of consent, subject refusal, physician decision, or death.
- Placebo and Pembrolizumab (PBO + PBZ): Participant received placebo tablets (identically matching in appearance to CC-486) administered orally daily on Days 1-14 plus pembrolizumab 200 mg administered as a 30-minute IV infusion on Day 1 of each 21-day cycle until radiologic disease progression, unacceptable toxicity, initiation of a new anticancer therapy, withdrawal of consent, subject refusal, physician decision, or death.
Period: Treatment Period
Arm/Group | CC-486 and Pembrolizumab (CC-486 + PBZ) | Placebo and Pembrolizumab (PBO + PBZ)
Started | 51 | 49
Completed (Completed = Not applicable according to the study design) | 0 | 0
Not Completed | 51 | 49
Not completed — Progressive Disease | 20 | 22
Not completed — Adverse Event | 14 | 6
Not completed — Symptomatic Deterioration | 4 | 3
Not completed — Death | 3 | 4
Not completed — Physician Decision | 1 | 2
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Non-compliance with Study Drug | 0 | 1
Not completed — Study Terminated by Sponsor | 0 | 1
Not completed — Miscellaneous | 7 | 9
Period: Survival Follow-Up Phase
Arm/Group | CC-486 and Pembrolizumab (CC-486 + PBZ) | Placebo and Pembrolizumab (PBO + PBZ)
Started | 36 | 35
Completed (Participants remained in follow-up until withdrawal of consent, death or lost to follow-up) | 0 | 0
Not Completed | 36 | 35
Not completed — Missing Status | 3 | 5
Not completed — Death | 18 | 12
Not completed — Alive | 13 | 16
Not completed — Lost to Follow-up | 2 | 2

BASELINE CHARACTERISTICS:
Population: The Intent-to-Treat (ITT) population includes all participants who were randomized, regardless of whether they received assigned treatment or not
Groups:
- Total: Total of all reporting groups
Arm/Group | CC-486 and Pembrolizumab (CC-486 + PBZ) | Placebo and Pembrolizumab (PBO + PBZ) | Total
Number analyzed (Participants) | 51 | 49 | 100
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: The Intent-to-Treat population includes all participants who were randomized.
  Years | 62.8 (10.03) | 64.9 (9.89) | 63.9 (9.96)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The Intent-to-Treat population includes all participants who were randomized.
  Participants
    Female | 25 | 18 | 43
    Male | 26 | 31 | 57
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: The Intent-to-Treat population includes all participants who were randomized.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 1 | 1
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 3 | 2 | 5
    White | 42 | 45 | 87
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 6 | 1 | 7
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — ECOG performance status is used by doctors and researchers to assess how a participant's disease is progressing, assess how the disease affects the daily living activities of the participant, and determine appropriate treatment and prognosis. 0 = Fully Active (Most Favorable Activity); 1 = Restricted activity but ambulatory; 2 = Ambulatory but unable to carry out work activities; 3 = Limited Self-Care; 4 = Completely Disabled, No self-care (Least Favorable Activity)
  Participants
    0 = Fully Active | 15 | 17 | 32
    1 = Restrictive but ambulatory | 36 | 32 | 68
    2 = ambulatory but unable to work | 0 | 0 | 0
    3 = limited self-care | 0 | 0 | 0
Stage at Primary Diagnosis [Count of Participants; unit: Participants] — Disease Stage means how big the tumor is and how far it has spread. Stages range from 0 (not spread) to IV (spread throughout the body). Stage 0 - the cancer has not spread beyond the inner lining of the lung Stage I - the cancer is small and hasn't spread to the lymph nodes Stage II - the cancer has spread to some lymph nodes near the original tumor Stage III - the cancer has spread to nearby tissue or spread to far away lymph nodes Stage IV - the cancer has spread to other organs of the body such as the other lung, brain, or liver.
  Participants
    Stage I | 3 | 2 | 5
    Stage II | 0 | 4 | 4
    Stage IIIA | 2 | 4 | 6
    Stage IIIB | 8 | 7 | 15
    Stage IV | 38 | 32 | 70
Histology [Count of Participants; unit: Participants] — The different types of lung cancer are described histologically by the types of cells the pathologist sees under the microscope. There are three major types of non-small cell lung cancer:
  Adenocarcinoma Squamous cell lung cancer (also called epidermoid carcinoma) Large cell lung cancer (Other)
  Participants
    Squamous cell carcinoma | 10 | 8 | 18
    Adenocarcinoma | 38 | 36 | 74
    Other | 3 | 5 | 8
Number of Metastatic Sites [Mean (Standard Deviation); unit: Metastatic sites] | 3.1 (1.33) | 2.8 (1.25) | 3.0 (1.29)
Number of Participants Randomized by Strata [Count of Participants; unit: Participants]
  Squamous Cell Carcinoma | 9 | 9 | 18
  Non-Squamous Cell Carcinoma | 42 | 40 | 82

OUTCOME MEASURES:

1. Primary Outcome: Kaplan Meier Estimate of Progression-Free Survival (PFS) Based on Food and Drug Administration (FDA) Methodology
Description: PFS was defined according to the FDA Methodology as the time in months from the date of randomization to the date of disease progression according to Response Evaluation Criteria In Solid Tumors (RECIST) Version 1.1 (documented by computed tomography scan, not including symptomatic deterioration) or death for (any cause) on or prior to the clinical cutoff date, whichever occurred earlier. Those who did not have disease progression or had not died as of the data cutoff date were censored at the time of the last radiologic assessment where the participant was documented to be progression-free prior to the data cutoff date. Progressive disease includes at least a 20% increase in the sum of diameters of target lesions from nadir or appearance of a new lesion.
Time Frame: From Day 1 of study drug treatment to the date of disease progression; up to the clinical cut-off date of 12 April 2017; overall maximum treatment duration was 61 weeks for the CC-486 + PBZ arm and 60 weeks for the PBZ + Placebo arm
Population: The Intent-to-Treat population includes all participants who were randomized, regardless of whether they received assigned treatment or not.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | CC-486 and Pembrolizumab (CC-486 + PBZ) | Placebo and Pembrolizumab (PBO + PBZ)
Number analyzed (Participants) | 51 | 49
months | 2.9 [1.8 to 4.0] | 4.0 [1.5 to 8.0]
Statistical Analysis 1: Comparison: CC-486 and Pembrolizumab (CC-486 + PBZ) vs Placebo and Pembrolizumab (PBO + PBZ); Test type: Superiority; p = 0.1789, Stratified Log-Rank Test; Stratified by squamous cell carcinoma versus non-squamous cell carcinoma; Hazard Ratio (HR) = 1.374, 90% CI 2-sided [0.926 to 2.038] — Hazard ratio and associated 2-sided 90% CIs were estimated using a Cox proportional hazard model

2. Secondary Outcome: Percentage of Participants Who Achieved a Complete Response (CR), Partial Response (PR) or Stable Disease (SD) for a Minimum Duration of 18 Weeks Compared to Baseline
Description: Disease control rate was defined as the percentage of participants who had confirmed stable disease, complete or partial response during the course of study, according to RECIST v1.1, as evaluated by the investigator.
  RECIST v 1.1 is defined as:
  * Complete response: disappearance of all target lesions
  * Partial response: at least a 30% decrease in the sum of diameters of target lesions from baseline
  * Stable disease: neither sufficient shrinkage to qualify for PR nor sufficient increase of lesions to qualify for progressive disease
  * Progressive Disease (PD): at least a 20% increase in the sum of diameters of target lesions from nadir or appearance of a new lesion. When stable disease was believed to be the best response, it must have met the minimum duration of 10 weeks from randomization.
Time Frame: Response was assessed every 6 weeks for the first 24 weeks, then every 9 weeks until DP, new anticancer initiation, or withdrawal of consent; maximum treatment exposure for CC-486 + PBZ was 61 weeks and 60 weeks for PBO +PBZ
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Arm/Group | CC-486 and Pembrolizumab (CC-486 + PBZ) | Placebo and Pembrolizumab (PBO + PBZ)
Number analyzed (Participants) | 51 | 49
Percentage of Participants | 25.5 [15.8 to 37.4] | 38.8 [27.1 to 51.5]
Statistical Analysis 1: Comparison: CC-486 and Pembrolizumab (CC-486 + PBZ) vs Placebo and Pembrolizumab (PBO + PBZ); Test type: Superiority; p = 0.1572, Cochran-Mantel-Haenszel; Stratified by squamous cell carcinoma vs non-squamous cell carcinoma; Disease Control Rate Difference = -13.3, 90% CI 2-sided [-29.0 to 3.5]

3. Secondary Outcome: Kaplan Meier Estimate of Overall Survival
Description: Overall survival (OS) was defined as the time in months between day 1 of treatment and death from any cause. Participants who were still alive as of the clinical cut-off date had their OS censored at the date of last contact or clinical cut-off, whichever was earlier. Participants who were lost to follow-up prior to the end of the study or who were withdrawn from the study were censored at the time of last contact.
Time Frame: From Day 1 of treatment up to the clinical cut-off date of 12 April 2017, whichever occurred earlier; median follow-up time for OS was 11.3 months in the CC-486 + PBZ arm and 12.2 months in the PBZ + Placebo arm
Population: The Intent-to-Treat population includes all participants who were randomized.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | CC-486 and Pembrolizumab (CC-486 + PBZ) | Placebo and Pembrolizumab (PBO + PBZ)
Number analyzed (Participants) | 51 | 49
months | 11.9 [7.2 to NA] — The upper limit was not estimable as participants were still alive at the time of the clinical cut-off date | NA [11.0 to NA] — Not estimable as participants were still alive at the time of the clinical cut-off date.
Statistical Analysis 1: Comparison: CC-486 and Pembrolizumab (CC-486 + PBZ) vs Placebo and Pembrolizumab (PBO + PBZ); Test type: Superiority; p = 0.2968, Stratified Log Rank; Stratified by squamous cell carcinoma vs non-squamous cell carcinoma); Hazard Ratio (HR) = 1.375, 90% CI 2-sided [0.830 to 2.276] — Hazard ratio and associated 2-sided 90% CIs were estimated using Cox proportional hazard model

4. Secondary Outcome: Percentage of Participants Who Achieved a Best Overall Response of Complete Response or Partial Response
Description: The best overall response is defined as the percentage of participants who achieved an objective confirmed complete response or partial response according to RECIST v1.1, compared with baseline where baseline was the last computed tomography (CT) scan obtained prior to or on day 1 of study treatment.
  RECIST v1.1 is defined as:
  * Complete response: disappearance of all target lesions
  * Partial response: at least a 30% decrease in the sum of diameters of target lesions from baseline
  * Stable disease: neither sufficient shrinkage to qualify for PR nor sufficient increase of lesions to qualify for progressive disease
  * Progressive Disease (PD): at least a 20% increase in the sum of diameters of target lesions from nadir or appearance of a new lesion.
Time Frame: Response was assessed every 6 weeks for the first 24 weeks, then every 9 weeks until DP, new anticancer initiation, or withdrawal of consent; maximum treatment exposure for CC-486 + PBZ was 61 weeks and 60 weeks for PBZ + PBO
Population: The Intent-to-Treat population includes all participants who were randomized.
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Arm/Group | CC-486 and Pembrolizumab (CC-486 + PBZ) | Placebo and Pembrolizumab (PBO + PBZ)
Number analyzed (Participants) | 51 | 49
Percentage of Participants | 19.6 [11.0 to 31.0] | 14.3 [6.9 to 25.2]
Statistical Analysis 1: Comparison: CC-486 and Pembrolizumab (CC-486 + PBZ) vs Placebo and Pembrolizumab (PBO + PBZ); Test type: Superiority; Overall Response Rate (ORR) Difference = 5.3, 90% CI 2-sided [-11.5 to 21.3] — The 90% exact unconditional confidence interval was used for ORR difference

5. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events
Description: Treatment-emergent adverse events (TEAEs) were defined as any adverse event (AE) or serious adverse event (SAE) that occurred or worsened on or after the day of the first dose of the investigational product (IP) through 28 days after the last dose of IP. In addition, any SAE with an onset date more than 28 day after the last dose of IP that was assessed by the investigator as related to IP was considered a TEAE. The severity of AEs was graded based on National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE), Version 4.0 and based on the following scale: Grade 1 = Mild; Grade 2 = Moderate Grade 3 = Severe Grade 4 = Life threatening Grade 5 = Death.
Time Frame: From date of first dose of study treatment until 30 days after the last dose of IP; overall maximum treatment duration was 61 weeks for the CC-486 + PBZ arm and 60 weeks for the PBZ + Placebo arm
Population: The safety population includes all participants who were randomized and received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | CC-486 and Pembrolizumab (CC-486 + PBZ) | Placebo and Pembrolizumab (PBO + PBZ)
Number analyzed (Participants) | 51 | 49
Participants
  Any TEAE | 51 | 49
  Any TEAE Related to Study Drug | 47 | 37
  Any Serious TEAE | 31 | 27
  Any Serious TEAE Related to Study Drug | 12 | 6
  Any CTC Grade 3/4 TEAE | 40 | 27
  Any CTC Grade 3/4 TEAE Related to Study Drug | 25 | 10
  Any TEAE Leading to Death | 6 | 9
  Any TEAE Leading to Dose Reduction | 10 | 1
  Any TEAE Leading to Dose Interruption | 32 | 20
  Any TEAE Leading to Drug Discontinuation | 20 | 8

6. Primary Outcome: Kaplan Meier Estimate of Progression-Free Survival (PFS) Based on European Medicines Agency Methodology
Description: Progression-free survival was defined according to EMA methodology as the time from the date of randomization to the date of disease progression according to Response Evaluation Criteria In Solid Tumors (RECIST) Version 1.1 (documented by computed tomography scan result, not including symptomatic deterioration) or death for (any cause) on or prior to the data cutoff date, whichever occurred earlier. Participants who did not have disease progression or had not died were censored at the last known time that the participant was progression free. However, occasional missing observations or initiation of subsequent new anticancer therapy would not result in censoring for this analysis. Progressive disease is at least a 20% increase in the sum of diameters of target lesions from nadir or appearance of a new lesion.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | CC-486 and Pembrolizumab (CC-486 + PBZ) | Placebo and Pembrolizumab (PBO + PBZ)
Number analyzed (Participants) | 51 | 49
months | 2.9 [1.8 to 4.0] | 4.0 [1.5 to 7.0]
Statistical Analysis 1: Comparison: CC-486 and Pembrolizumab (CC-486 + PBZ) vs Placebo and Pembrolizumab (PBO + PBZ); Test type: Superiority; p = 0.1990, Stratified Log-Rank Test; Stratified by squamous cell carcinoma versus non-squamous cell carcinoma; Hazard Ratio (HR) = 1.352, 90% CI 2-sided [0.914 to 2.000] — Hazard ratio and associated 2-sided 90% CIs were estimated using a Cox proportional hazard model

7. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to Infinity (AUC∞) of CC-486
Description: Area under the plasma concentration-time curve from Time 0 extrapolated to infinity, calculated as [AUCt + Ct/ λz]. Ct is the last quantifiable concentration. No AUC extrapolation was performed with unreliable λz. If AUC % extrap is ≥25%, AUCi inf was not reported.
Time Frame: Pharmacokinetic (PK) blood samples collected at 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6 and 8 hours after CC-486 administration on Cycle 1 Day 1 and Cycle 2 Day 1
Population: The PK population includes participants with evaluable CC-486 plasma PK profile.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | CC-486 and Pembrolizumab (CC-486 + PBZ)
Number analyzed (Participants) | 15
ng*h/mL
  Cycle 1 Day 1 | 156.0 (82.64)
  Cycle 2 Day 1: number analyzed (Participants) | 13
  Cycle 2 Day 1 | 212.7 (78.06)

8. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to the Last Measurable Concentration (AUCt) of CC-486
Description: Area under the plasma concentration-time curve from Time 0 to the time of the last quantifiable concentration, calculated by linear trapezoidal method when concentrations are increasing and the logarithmic trapezoidal method when concentrations are decreasing.
Time Frame: PK blood samples collected at 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6 and 8 hours after CC-486 administration on Cycle 1 Day 1 and Cycle 2 Day 1
Population: The PK population includes participants with evaluable CC-486 plasma PK profile.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng·h/mL
Arm/Group | CC-486 and Pembrolizumab (CC-486 + PBZ)
Number analyzed (Participants) | 15
ng·h/mL
  Cycle 1 Day 1 | 152.3 (85.67)
  Cycle 2 Day 1: number analyzed (Participants) | 14
  Cycle 2 Day 1 | 196.6 (88.63)

9. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of CC-486
Description: Maximum observed plasma concentration, obtained directly from the observed concentration versus time data.
Time Frame: as for outcome 8
Population: The PK population includes participants with evaluable CC-486 plasma PK profile.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | CC-486 and Pembrolizumab (CC-486 + PBZ)
Number analyzed (Participants) | 15
ng/mL
  Cycle 1 Day 1 | 94.7 (69.49)
  Cycle 2 Day 1: number analyzed (Participants) | 14
  Cycle 2 Day 1 | 110.0 (73.46)

10. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) of CC-486
Description: Time to maximum observed plasma concentration obtained directly from the observed concentration versus time data.
Time Frame: as for outcome 8
Population: The PK population includes participants with evaluable CC-486 plasma PK profile.
Measure: Median (Full Range); unit: hours
Arm/Group | CC-486 and Pembrolizumab (CC-486 + PBZ)
Number analyzed (Participants) | 15
hours
  Cycle 1 Day 1 | 1.5 [0.5 to 3.0]
  Cycle 2 Day 1: number analyzed (Participants) | 14
  Cycle 2 Day 1 | 1.5 [0.5 to 3.5]

11. Secondary Outcome: Terminal Phase of Half-life (T1/2) of CC-486
Description: Terminal phase half-life in plasma, calculated as [(ln 2)/λz]. t1/2 was only be calculated when a reliable estimate for λz could be obtained.
Time Frame: as for outcome 8
Population: The PK population includes participants with evaluable CC-486 plasma PK profile.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | CC-486 and Pembrolizumab (CC-486 + PBZ)
Number analyzed (Participants) | 15
hours
  Cycle 1 Day 1 | 0.7 (30.22)
  Cycle 2 Day 1: number analyzed (Participants) | 13
  Cycle 2 Day 1 | 0.9 (91.72)

12. Secondary Outcome: Apparent Total Plasma Clearance (CL/F) of CC-486
Description: Apparent total plasma clearance (CL/F) of CC-486 was calculated as Dose/AUC∞
Time Frame: as for outcome 8
Population: The PK population includes participants with evaluable CC-486 plasma PK profile.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters/hour
Arm/Group | CC-486 and Pembrolizumab (CC-486 + PBZ)
Number analyzed (Participants) | 15
Liters/hour
  Cycle 1 Day 1 | 1922.7 (82.64)
  Cycle 2 Day 1: number analyzed (Participants) | 13
  Cycle 2 Day 1 | 1410.4 (78.06)

13. Secondary Outcome: Apparent Volume of Distribution (Vd/F) of CC-486
Description: Apparent volume of distribution, was calculated according to the equation: Vd/F = (CL/F)/λz
Time Frame: as for outcome 8
Population: The PK population includes participants with evaluable CC-486 plasma PK profile.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | CC-486 and Pembrolizumab (CC-486 + PBZ)
Number analyzed (Participants) | 15
Liters
  Cycle 1 Day 1 | 1836.2 (100.80)
  Cycle 2 Day 1: number analyzed (Participants) | 13
  Cycle 2 Day 1 | 1777.1 (163.62)

ADVERSE EVENTS:
Time Frame: From date of first dose of study treatment until 30 days after the last dose of IP; overall maximum treatment duration was 61 weeks for the CC-486 + PBZ arm and 60 weeks for the for the PBZ + PBO arm.
Description: All-cause mortality timeframe includes deaths from day 1 of study treatment to final data cut-off date of 12 April 2017
Groups:
- CC-486+Pembrolizumab: Participants received CC-486 300 mg tablets by mouth (PO) on Days 1-14 of each 21-day treatment cycle and pembrolizumab (PBZ) 200 mg administered as a 30-minute intravenous (IV) infusion on Day 1 of each 21-day cycle until radiologic disease progression (DP), unacceptable toxicity, initiation of a new anticancer therapy, withdrawal of consent, subject refusal, physician decision, or death.
- Pembrolizumab+Placebo: Participants received placebo tablets orally on days 1-14 plus pembrolizumab 200 mg administered as a 30-minute IV infusion on day 1 of a 21-day cycle until radiologic disease progression, unacceptable toxicity, initiation of a new anticancer therapy, withdrawal of consent, subject refusal, physician decision, or death.
Arm/Group | CC-486+Pembrolizumab | Pembrolizumab+Placebo
All-Cause Mortality (participants affected / at risk) | 23/51 | 20/49
Serious Adverse Events (participants affected / at risk) | 31/51 | 27/49
Other Adverse Events (participants affected / at risk) | 51/51 | 48/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CC-486+Pembrolizumab (N=51) | Pembrolizumab+Placebo (N=49)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0
Diplopia (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 4 | 0
Vomiting (Gastrointestinal disorders) | 4 | 0
Asthenia (General disorders) | 1 | 0
Death (General disorders) | 0 | 1
Fatigue (General disorders) | 1 | 0
General physical health deterioration (General disorders) | 3 | 1
Non-cardiac chest pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 3
Autoimmune hepatitis (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 2 | 1
Hepatitis toxic (Hepatobiliary disorders) | 1 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 1
Device related infection (Infections and infestations) | 1 | 0
Intervertebral discitis (Infections and infestations) | 1 | 0
Lower respiratory tract infection bacterial (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 4
Respiratory tract infection (Infections and infestations) | 1 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0
Drug administration error (Injury, poisoning and procedural complications) | 1 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ataxia (Nervous system disorders) | 0 | 1
Dysarthria (Nervous system disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 0 | 1
Irritability (Psychiatric disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Nephritis (Renal and urinary disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CC-486+Pembrolizumab (N=51) | Pembrolizumab+Placebo (N=49)
Anaemia (Blood and lymphatic system disorders) | 12 | 8
Leukopenia (Blood and lymphatic system disorders) | 3 | 1
Neutropenia (Blood and lymphatic system disorders) | 8 | 1
Tachycardia (Cardiac disorders) | 3 | 0
Hyperthyroidism (Endocrine disorders) | 2 | 3
Hypothyroidism (Endocrine disorders) | 3 | 3
Abdominal pain (Gastrointestinal disorders) | 8 | 4
Abdominal pain upper (Gastrointestinal disorders) | 5 | 2
Constipation (Gastrointestinal disorders) | 18 | 9
Diarrhoea (Gastrointestinal disorders) | 20 | 12
Dyspepsia (Gastrointestinal disorders) | 4 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 1
Nausea (Gastrointestinal disorders) | 37 | 13
Stomatitis (Gastrointestinal disorders) | 4 | 1
Vomiting (Gastrointestinal disorders) | 32 | 9
Asthenia (General disorders) | 22 | 17
Fatigue (General disorders) | 10 | 3
General physical health deterioration (General disorders) | 3 | 1
Non-cardiac chest pain (General disorders) | 4 | 0
Oedema peripheral (General disorders) | 5 | 8
Pyrexia (General disorders) | 18 | 13
Hypertransaminasaemia (Hepatobiliary disorders) | 3 | 0
Bronchitis (Infections and infestations) | 0 | 5
Oral candidiasis (Infections and infestations) | 3 | 0
Upper respiratory tract infection (Infections and infestations) | 5 | 2
Alanine aminotransferase increased (Investigations) | 4 | 2
Aspartate aminotransferase increased (Investigations) | 4 | 3
Blood alkaline phosphatase increased (Investigations) | 4 | 0
Weight decreased (Investigations) | 11 | 3
Decreased appetite (Metabolism and nutrition disorders) | 19 | 20
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 6 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 6 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 4
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 5
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 5
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 8
Dizziness (Nervous system disorders) | 5 | 4
Headache (Nervous system disorders) | 5 | 4
Paraesthesia (Nervous system disorders) | 3 | 4
Somnolence (Nervous system disorders) | 2 | 3
Anxiety (Psychiatric disorders) | 4 | 2
Insomnia (Psychiatric disorders) | 3 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 12 | 17
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 | 11
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 4
Rash pruritic (Skin and subcutaneous tissue disorders) | 4 | 2
Hypertension (Vascular disorders) | 6 | 1
Hypotension (Vascular disorders) | 4 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Results from a center cannot be submitted for publication before results of multicenter study are published unless it is more than 1 year from study completion. Investigator can publish if manuscript is submitted to Celgene 60 days prior to submission. If Celgene decides publication would hinder drug development, Investigator must delay submission for up to 90 additional days. Investigator must delete confidential information before submission or defer publication to permit patent applications.

DOCUMENTS (3):
  • Study Protocol: CC-486-NSCL-001_original protocol_Redacted.15May2015 (2015-05-15): https://cdn.clinicaltrials.gov/large-docs/86/NCT02546986/Prot_000.pdf
  • Study Protocol: CC-486-NSCL-001.ProtocolAM1.14December 2015 (2015-12-14): https://cdn.clinicaltrials.gov/large-docs/86/NCT02546986/Prot_001.pdf
  • Statistical Analysis Plan (2017-06-28): https://cdn.clinicaltrials.gov/large-docs/86/NCT02546986/SAP_002.pdf